CLINICAL TRIAL: NCT07206576
Title: Acute Effects of Percussion Massage Therapy on Balance, Explosive Power, and Functional Performance in Adolescent Cyclists: A Randomized Controlled Trial
Brief Title: Acute Effects of Percussion Massage Therapy in Adolescent Cyclists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Emre DANSUK, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-6304
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Balanced
Keywords: Cycling; Functional performance; Explosive strength; Balance; Vibration therapy

STUDY DESIGN:
Intervention Model Description: This study is designed as a two-arm, parallel-group, randomized controlled trial. A total of 32 adolescent competitive cyclists aged 12-15 years will be randomly assigned (1:1 ratio) to either the intervention group receiving percussion massage therapy (PMT) or the control group undergoing passive rest.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percussion Massage Therapy Group (Experimental): Participants in this group will receive a single session of percussion massage therapy (PMT) using the Compex® Fixx™ 2.0 device applied bilaterally to the gluteus maximus, quadriceps femoris, and gastrocnemius muscles for 3 minutes per muscle group at 41.7 Hz.
  Interventions: Device: a percussion massage gun
- Control Group (No Intervention): Participants in this group will not receive any intervention. They will remain seated in a resting position for an equivalent duration (approximately 18 minutes) to match the intervention group's time frame.

INTERVENTIONS:
Device: a percussion massage gun — Participants assigned to the intervention group will receive a single session of percussion massage therapy (PMT) using the Compex® Fixx™ 2.0 handheld device. The treatment will be applied bilaterally to three major muscle groups: gluteus maximus, quadriceps femoris, and gastrocnemius.
  The device will operate at a high intensity setting (Level 4) with a frequency of 41.7 Hz.
  A wedge-shaped applicator head will be used to ensure consistent pressure across the treatment area.
  Each muscle group will be treated for 3 minutes, following a standardized linear stroke pattern from proximal to distal and back.
  The total duration of the intervention will be approximately 18 minutes.
  The intervention will be performed once, immediately before the post-test evaluations, and aims to assess acute effects on neuromuscular performance.
  Arms: Percussion Massage Therapy Group

SUMMARY:
This randomized controlled trial aims to investigate the acute effects of percussion massage therapy (PMT) on balance, explosive strength, and functional performance in adolescent competitive cyclists aged 12-15. A total of 32 participants will be randomly assigned to either a PMT group, which will receive a single session of vibration-based therapy using a handheld percussion device (Compex Fixx 2.0), or a control group with passive rest. Performance parameters will be assessed using the Y Balance Test, vertical jump, hop tests, 10-second sprint cycling, and isometric muscle strength via dynamometry. The study seeks to determine whether PMT offers short-term neuromuscular benefits that may enhance cycling performance in youth athletes.

DETAILED DESCRIPTION:
Cycling is a sport that requires repetitive and rhythmic activation of the lower extremity muscles, where balance, endurance, and muscular power are critical. In adolescent athletes aged 12-15, musculoskeletal structures are still developing, and interventions aimed at enhancing performance must be carefully investigated in terms of both efficacy and safety.

Percussion massage therapy (PMT) is a novel method that combines elements of traditional massage and vibration therapy, applying rapid mechanical pulses to soft tissues using handheld devices. PMT has gained popularity in recent years due to its potential to enhance circulation, reduce muscle stiffness, and improve neuromuscular function. Studies suggest that PMT can produce acute effects such as improved proprioception, reduced muscle tone, and enhanced explosive performance.

This randomized controlled trial aims to evaluate the acute effects of PMT on dynamic balance, explosive strength, and functional performance in young competitive cyclists. Thirty-two participants, aged 12 to 15, who have been licensed cyclists for at least 2 years and train regularly, will be randomly assigned to either an intervention group receiving PMT or a control group undergoing passive rest.

The intervention group will receive a single session of PMT using the Compex® Fixx™ 2.0 device, applied bilaterally to the gluteus maximus, quadriceps femoris, and gastrocnemius muscles at 41.7 Hz for 3 minutes per muscle group. The control group will remain seated for an equivalent rest period.

Performance outcomes will be assessed using the Y Balance Test, Vertical Jump Test, single-leg hop test (triple hop), 10-second cycling sprint test, and handheld dynamometry to measure isometric muscle strength. In addition, subjective muscle relaxation will be evaluated pre- and post-intervention using the Numeric Rating Scale (NRS).

The findings of this study will contribute to the limited body of evidence regarding vibration-based interventions in youth athletes and help determine whether PMT is a viable strategy to acutely improve neuromuscular performance in adolescent cyclists.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 12 and 15 years
* Licensed competitive cyclist for at least 2 years
* Participating in at least 4 training sessions per week
* No lower extremity injuries in the past 6 months
* Voluntary participation by signing the informed consent form

Exclusion Criteria:

* History of surgery in the knee, hip, or ankle joints
* Presence of neurological, vestibular, or systemic balance disorders
* Use of medications that may affect performance
* Any orthopedic condition that prevents participation in performance tests

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2025-09-30 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Y Balance Test Composite Score | Pre-intervention and immediately post-intervention
  The Y Balance Test will be used to assess dynamic balance by measuring reach distances in three directions (anterior, posteromedial, and posterolateral) while standing on one leg. Each direction will be tested three times, and the average reach distance will be normalized to leg length. A composite score will be calculated and expressed as a percentage to evaluate overall dynamic balance capacity. Higher scores indicate better balance performance.

SECONDARY OUTCOMES:
Single-Leg Hop Distance (Triple Hop Test) | Pre-intervention and immediately post-intervention
  The Triple Hop Test evaluates lower limb strength, power, and dynamic stability. Participants will perform three consecutive forward hops on the same leg along a straight line, aiming for maximal distance. The total distance from toe-off to the final landing point will be measured in centimeters. The longest of three valid trials will be recorded. Increased hop distance indicates improved functional performance.
Isometric Muscle Strength (Gluteus Maximus, Quadriceps, Gastrocnemius) | Pre-intervention and immediately post-intervention
  Isometric strength of gluteus maximus, quadriceps femoris, and gastrocnemius will be measured using a handheld dynamometer. Standardized positioning and stabilization techniques will be used to ensure reliability. Three maximal contractions will be performed for each muscle, and the highest value (in Newtons) will be recorded for analysis. Greater force output reflects improved neuromuscular capacity.
Peak Power Output | Pre-intervention and immediately post-intervention
  Sprint cycling performance will be assessed using a stationary cycle ergometer. After a warm-up, participants will perform a 10-second all-out sprint with standardized resistance. Peak power (Watts) will be recorded as an indicator of anaerobic capacity.
Sprint Distance | Pre-intervention and immediately post-intervention
  During the same 10-second sprint test, the total distance covered (meters) will be recorded as an indicator of explosive leg power.
Subjective Muscle Relaxation (Numeric Rating Scale - NRS) | Pre-intervention and immediately post-intervention
  Subjective perception of muscle relaxation will be assessed using the Numeric Rating Scale (NRS), ranging from 0 (no relaxation) to 10 (complete relaxation). Participants will rate their perceived muscle tension and relaxation immediately before and after the intervention to quantify perceived benefits.

CONTACTS AND LOCATIONS:
Locations (1):
- Tayfun Arslan, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No